CLINICAL TRIAL: NCT01719692
Title: Prospective Multi-center Randomized Controlled Low-dose Rituximab Regimens in Chinese Adult Patients With Immune Thrombocytopenia
Brief Title: Low-dose Rituximab Regimens in Chinese Adult Patients With Immune Thrombocytopenia
Acronym: ITP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Langfang Traditional Chinese Medicine Hospital (Unknown); Henan Cancer Hospital (Other Government); The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2012001
Record Dates: First submitted 2012-10-26; First posted 2012-11-01 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2024-03

CONDITIONS: Immune Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab A group (Experimental): 375mg/m2 for once
  Interventions: Drug: Rituximab
- Rituximab B group (Active Comparator): 100mg/week for four weeks
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab
  Other Names: Trade names Rituxan and MabThera

SUMMARY:
A comparative study with rituximab (100 mg weekly for 4 weeks and 375mg/m2 for once) shows low dose rituximab may be a useful alternative therapy in patients with ITP.The aim of this study is to compare the efficacy and tolerability of two different regimens of low doses rituximab for the treatment of adult patients with ITP.

DETAILED DESCRIPTION:
This is a multicentre, prospective, open-label, randomised controlled trial. The aim of this study will compare the long-term efficacy and safety of two low-dose rituximab regimens in adult Chinese patients with glucocorticoid-resistant/dependent or relapsed ITP. Group A will receive rituximab100 mg weekly for four weeks, and group B will receive rituximab 375 mg/m2 once. After initiating treatment, if the patient has at least two consecutive evaluations (interval >7 days) without rescue therapy and a platelet count >50×109/L, the concomitant medications such as glucocorticoids can be reduced or stopped.

Within 3 months of the last rituximab dose, rescue therapy is recommended if the patient has an extremely low platelet count and an obvious bleeding tendency. Rescue therapy is limited to IVIG (0.4 g/kg per day for 3-5 days) and glucocorticoid (methylprednisolone 0.8 mg/kg per day for 7-14 days or equivalent dose of other glucocorticoids).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old;
* Diagnosis of primary immune thrombocytopenia according to the guidelines of American Society of Hematology for at least 3 months before inclusion;
* Platelet count <30×109/L (measured at least twice during the screening, with at least a 1-week interval);
* Failed or dependent on or relapsed after previous treatment with glucocorticoid;
* If on glucocorticoid maintenance therapy, dose ≤0.5 mg/kg prednisone or equivalent and stabilised for at least 4 weeks;
* Drugs such as azathioprine, danazol, cyclosporine A, tacrolimus, and sirolimus stopped for at least 4 weeks;
* Splenectomy more than 6 months previously;
* Previous rescue therapy of ITP (including methylprednisolone, platelet transfusion and IVIG) completed at least 2 weeks before the first administration;
* Liver and kidney function (including alanine aminotransferase, aspartate aminotransferase, total bilirubin, serum creatine, urea nitrogen, etc.) less than 1.5 times the upper limit of normal value;
* Eastern Cooperative Oncology Group performance status ≤2;
* Cardiac function classification (New York Heart Association) ≤2;
* Understand the research procedure and voluntarily sign a written informed consent form.

Exclusion Criteria:

* Patients with secondary thrombocytopenia (including myelodysplastic syndrome, aplastic anemia, common variant immunodeficiency disease, hereditary thrombocytopenia, drug-induced thrombocytopenia, pseudothrombocytopenia, connective tissue disease secondary thrombocytopenia, thrombocytopenia after liver disease, etc.);
* Previous treatment of RTX or allergic to RTX;
* Uncontrollable primary diseases of important organs (including malignant tumor, liver failure, heart failure, kidney failure and other diseases);
* HIV-positive status;
* Active infection including hepatitis B (HBV), hepatitis C (HCV) and other viral antigens or DNA, RNA positive; cytomegalovirus, Epstein-Barr virus, syphilis chronic or active infection. If HBV core antibodies are positive, HBV-DNA testing is required.
* Extensive and severe bleeding, such as hemoptysis, upper gastrointestinal hemorrhage, intracranial hemorrhage, etc.
* Heart disease or arrhythmia need treatment, or poorly controlled hypertension;
* Thrombotic diseases including pulmonary embolism, thrombosis, atherosclerosis, etc.;
* Previously allogeneic stem cell transplantation or organ transplantation;
* Mental disorders who are unable to obtain informed consent normally and participate in trials and follow-up;
* Symptoms of toxicity from pre-trial treatment have not resolved;
* Other severe conditions that may limit participation in the trial (e.g., diabetes; severe cardiac insufficiency; myocardial infarction or unstable arrhythmia or unstable angina within the last 6 months; gastric ulcer; active autoimmune diseases, etc.);
* Sepsis or other irregular bleeding;
* Taking antiplatelet drugs;
* pregnancy, suspected pregnancy (urine human chorionic gonadotropin positive during screening) or lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Overall response rate at week 12 | Patients will be followed for 6 months at least after Rituximab treatment.
  Overall response rate was defined as proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least twice the baseline platelet count without bleeding and subjects with a platelet count ≥ 100 × 10^9/L without bleeding at week 12 after initial administration in absence of rescue therapy, and without having had dose increment of corticosteroids during the study period.

SECONDARY OUTCOMES:
Sustained response rate over 6 months and 1, 2, 3, 4, and 5 years after RTX initiation | Patients will be followed for 6 months at least after Rituximab treatment.
  Proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least twice the baseline platelet count without bleeding and subjects with a platelet count ≥ 100 × 10^9/L without bleeding at 6 months and 1, 2, 3, 4, and 5 years after initial administration in absence of rescue therapy
Time to response (TTR) | 6 months
  Time needed from treatment initiation to platelet count ≥30×10^9/L and at least twice the baseline platelet count.
Number of subjects with clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale | 3 months
  Changes of the subjects' numbers in WHO bleeding score after RTX treatment according to the reported World Health Organization's Bleeding Scale at month 3. The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Adverse events assessment | 12 months
  Incidence, severity, and relationship of treatment emergent adverse events during the study period

CONTACTS AND LOCATIONS:
Overall Officials: RENCHI YANG, Dr, Principal Investigator — Hospital of Blood disease
Locations (1):
- Hospital of Blood disease, Tianjin, Tianjin Municipality, China